CLINICAL TRIAL: NCT04663360
Title: Medication Monitoring in General Practice: Clinical Impact of Implementing a Nurse-led Adverse Drug Reaction (ADRe) Profile in Older Adults With 5 or More Prescribed Medicines
Brief Title: Medication Monitoring for Older Adults in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swansea University (Other)
Collaborators: Abertawe Bro Morgannwg University Health Board (Other); Hywel Dda Health Board (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Swansea Nursing
Record Dates: First submitted 2020-11-26; First posted 2020-12-11 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2020-11

CONDITIONS: Polypharmacy
Keywords: medicines management; adverse drug reaction; nurses; primary care
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Intervention Model Description: Participating GP practices will be randomised into an intervention and control arms.
Masking Description: Masking is not possible due to cluster randomisation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention to be administered: Adverse Drug Reactions (ADRe) Profile. asks nurses to systematically check patients for the manifestation of itemised adverse side effects or undesirable effects of their primary care medicines, as listed in the BNF and manufacturers' Summaries of Product Characteristics (SmPCs), and seminal texts documenting known ADRs. Nurses are asked to share the identified problems with prescribers and pharmacists overseeing medicines charts.
  Interventions: Other: Adverse Drug Reaction (ADRe) Profile
- Control (No Intervention): Usual clinical care.

INTERVENTIONS:
Other: Adverse Drug Reaction (ADRe) Profile — ADRe asks nurses to systematically check patients for the manifestation of itemised adverse side effects or undesirable effects of their primary care medicines, as listed in the BNF and manufacturers' Summaries of Product Characteristics (SmPCs), and seminal texts documenting known ADRs. Nurses are asked to share the identified problems with prescribers and pharmacists overseeing medicines charts.
  Arms: Intervention

SUMMARY:
Polypharmacy has the potential to harm older adults by causing cognitive impairment, falls, and hospitalisations. Many adverse drug reactions could be prevented with closer monitoring. This project will establish the effectiveness of the nurse-led intervention - the ADRe Profile - for medicines commonly prescribed in primary care and evaluate intervention implementation in general practices.

DETAILED DESCRIPTION:
The number of medicines people take is increasing. Older adults are particularly at risk of adverse drug reactions due to polypharmacy. Adverse drug reactions cause avoidable patient harm, and around 5-8% of unplanned hospital admissions in the UK, costing the NHS £1.5-2.5bn pa. Many adverse drug reactions could be prevented with closer monitoring. The nurse-led Adverse Drug Reactions Profile (ADRe Profile) represents a unique instrument that records patients' observations and self-reported information on signs and symptoms that is likely to relate to an adverse reaction to medications. This project will establish the effectiveness of ADRe Profile in identifying patient problems possibly resulting from medicines in general practices and will be implemented in 3 phases.

Phase 1 (4 months) Validity and reliability testing of the ADRe Profile will be performed with key stakeholders (patients, nurses, care assistants, GP's and pharmacists), before introducing the tool to general practices. Feasibility testing will also be undertaken.

Phase 2 (12 months) The aim of this phase is to test whether the ADRe Profile identifies and ameliorates health problems. The practice nurse (or the researcher) will perform an ADRe consultation with a group of eligible service users and compare the number and nature of health and well-being problems identified with a similar group of service users who receive normal care.

Phase 3 (6 months) Finally, to further explore the impact of the ADRe Profile, the researchers will conduct semi-structured interviews with health professionals (nurses, care assistants, GPs and pharmacists) and service users.

The investigators hope that this study will help patients gain maximum benefits from their medicines and support nurses, pharmacists and GP's to reduce any bothersome side effects and problems that, if not addressed promptly, can lead to hospital admissions.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria:

Patients:

* age > 64 years
* with a long-term condition
* prescribed > 5 medications daily. (Vitamin and nutritional supplements and moisturising skin preparations will not be counted as 'medicines'.)
* Willing and able to give informed, signed consent themselves, or where capacity is lacking in the opinion of their nurses, a consultee/representative accompanying the patient who is willing to give advice and assent to the service user participating and sign on their behalf.

Exclusion Criteria:

Patients:

* Age < 64 years
* Without any long-term conditions
* Prescribed < 5 medications daily
* Not willing to participate
* Unable to consent and no consultee/representative present
* Not fluent in English or Welsh (unless a family member can assist with translation)
* Receiving palliative care
* Expected to remain in the practice for the next 12 months

Min Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-10-04 (Actual)

PRIMARY OUTCOMES:
Level of completion of all items in the video call-completed ADRe Profile | 4 months from the start of the study
  Comparison of completeness of the ADRe Profile completed through a video call with ADRe Profiles previously completed in person
Inter-rater reliability of patient versus nurse (or nurse-researcher) completed ADRe Profile (Cohen's Kappa). | 4 months from the start of the study
  To determine how much of the potential variability of the records is due to errors in measurement, to estimate a degree to which service users accurately evaluate their symptoms when compared with a nurse researcher. Cohen's Kappa will be calculated.
Calculated percentage and described nature of items on the ADRe Profile that can be populated from accessing the nursing and medical notes. | 16 months from the start of the study
  Establishing the overlap of information - the number and nature of the ADRe items that have previously been collected and recorded in the patients' nursing and medical notes.
Clinical impact on service users, including new problems identified (number and nature) and problems addressed (number and nature) | 16 months from the start of the study
  Number of patients with a change in signs and symptoms related to adverse effects of prescribed medicines. Care quality/ clinical gain/ benefit to patients as recorded in notes and on the Profile by the number and nature of all health problems addressed, particularly serious adverse events.
Prescription changes | 16 months from the start of the study
  Number of patients with changes in prescription regimens: drug or dose. Number and nature of changes.
Description of stakeholder views on ADRe Profile implementation effectiveness (survey rating of the ADRe Profile - Likert scale) | 22 months from the start of the study
  A brief survey will be distributed to the main stakeholders (patients, nurses, GP's and pharmacists) following completion of Randomised Controlled Trial.
Description of stakeholder views on ADRe Profile implementation feasibility (eliciting interview themes) | 22 months from the start of the study
  Semi-structured interview with the main stakeholders (patients, nurses, GP's and pharmacists) to explore their views on feasibility of ADRe Profile integration in GP practices.

SECONDARY OUTCOMES:
Calculation of the average nurses', GP's and pharmacists' length of time per one ADRe Profile completion | 16 months from the start of the study
  Average length of the health professionals' time involvement with one ADRe Profile
Calculation of the cost of nurses', GP's and pharmacists' time, based on average national salary cost per hour. | 16 months from the start of the study
  Estimated costs of ADRe implementation in GP practices
Description of the main stakeholders' views on multidisciplinary collaboration (eliciting interview themes) | 22 months from the start of the study
  Semi-structured interview with the main stakeholders (patients, nurses, GP's and pharmacists) to explore their views on whether and how ADRe Profile contributed to multidisciplinary collaboration between nurses, doctors and pharmacists
Description of the patients' views on the contribution of ADRe Profile to patient-centered care (eliciting interview themes). | 22 months from the start of the study
  Semi-structured interview with the patients to seek their views on whether and how ADRe Profile contributes to patient-centered care

CONTACTS AND LOCATIONS:
Overall Officials: Sue Jordan, PhD, Study Chair — Swansea University
Locations (1):
- Aneurin Bevan Health Board, Newport, Gwent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gabe ME, Murphy F, Davies GA, Russell IT, Jordan S. Medication monitoring in a nurse-led respiratory outpatient clinic: pragmatic randomised trial of the West Wales Adverse Drug Reaction Profile. PLoS One. 2014 May 5;9(5):e96682. doi: 10.1371/journal.pone.0096682. eCollection 2014. PMID 24798210
- [Background] Jones R, Moyle C, Jordan S. Nurse-led medicines monitoring: a study examining the effects of the West Wales Adverse Drug Reaction Profile. Nurs Stand. 2016 Nov 30;31(14):42-53. doi: 10.7748/ns.2016.e10447. PMID 27902153
- [Background] Jordan S. Managing adverse drug reactions: an orphan task. J Adv Nurs. 2002 Jun;38(5):437-48. doi: 10.1046/j.1365-2648.2002.02205.x. PMID 12028277
- [Background] Jordan S, Tunnicliffe C, Sykes A. Minimizing side-effects: the clinical impact of nurse-administered 'side-effect' checklists. J Adv Nurs. 2002 Jan;37(2):155-65. doi: 10.1046/j.1365-2648.2002.02064.x. PMID 11851783
- [Background] Jordan S, Gabe M, Newson L, Snelgrove S, Panes G, Picek A, Russell IT, Dennis M. Medication monitoring for people with dementia in care homes: the feasibility and clinical impact of nurse-led monitoring. ScientificWorldJournal. 2014 Feb 23;2014:843621. doi: 10.1155/2014/843621. eCollection 2014. PMID 24707218
- [Background] Jordan S, Gabe-Walters ME, Watkins A, Humphreys I, Newson L, Snelgrove S, Dennis MS. Nurse-Led Medicines' Monitoring for Patients with Dementia in Care Homes: A Pragmatic Cohort Stepped Wedge Cluster Randomised Trial. PLoS One. 2015 Oct 13;10(10):e0140203. doi: 10.1371/journal.pone.0140203. eCollection 2015. PMID 26461064
- [Background] Jordan S, Banner T, Gabe-Walters M, Mikhail JM, Panes G, Round J, Snelgrove S, Storey M, Hughes D; Medicines' Management Group, Swansea University. Nurse-led medicines' monitoring in care homes, implementing the Adverse Drug Reaction (ADRe) Profile improvement initiative for mental health medicines: An observational and interview study. PLoS One. 2019 Sep 11;14(9):e0220885. doi: 10.1371/journal.pone.0220885. eCollection 2019. PMID 31509537
- [Background] Mangoni AA, Jackson SH. Age-related changes in pharmacokinetics and pharmacodynamics: basic principles and practical applications. Br J Clin Pharmacol. 2004 Jan;57(1):6-14. doi: 10.1046/j.1365-2125.2003.02007.x. PMID 14678335
- [Background] Masnoon N, Shakib S, Kalisch-Ellett L, Caughey GE. What is polypharmacy? A systematic review of definitions. BMC Geriatr. 2017 Oct 10;17(1):230. doi: 10.1186/s12877-017-0621-2. PMID 29017448
- [Background] NHS Digital (2017). Health Survey for England 2016: Prescribed medicines. https://files.digital.nhs.uk/pdf/3/c/hse2016-pres-med.pdf
- [Background] NICE Medicines and Prescribing Centre. (2015). Medicines optimisation: the safe and effective use of medicines to enable the best possible outcomes. NICE Guideline 5. London: NICE
- [Background] Sirois C, Domingues NS, Laroche ML, Zongo A, Lunghi C, Guenette L, Kroger E, Emond V. Polypharmacy Definitions for Multimorbid Older Adults Need Stronger Foundations to Guide Research, Clinical Practice and Public Health. Pharmacy (Basel). 2019 Aug 29;7(3):126. doi: 10.3390/pharmacy7030126. PMID 31470621
- [Derived] Logan V, Hughes D, Turner A, Carter N, Jordan S. Breaking barriers: feasibility of a cluster randomised trial evaluating an instrument for identifying and ameliorating adverse drug reactions. BMJ Open. 2026 Jan 27;16(1):e099627. doi: 10.1136/bmjopen-2025-099627. PMID 41592836
- [Derived] Logan V, Carter N, Hughes D, Turner A, Jordan S. Reducing Adverse Drug Reactions for Older People in the Community: Evaluating the Validity and Reliability of the ADRe Profile. J Nurs Manag. 2025 May 14;2025:9921349. doi: 10.1155/jonm/9921349. eCollection 2025. PMID 40401039
- [Derived] Logan V, Bamsey A, Carter N, Hughes D, Turner A, Jordan S. Clinical Impact of Implementing a Nurse-Led Adverse Drug Reaction Profile in Older Adults Prescribed Multiple Medicines in UK Primary Care: A Study Protocol for a Cluster-Randomised Controlled Trial. Pharmacy (Basel). 2022 Apr 28;10(3):52. doi: 10.3390/pharmacy10030052. PMID 35645331

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT04663360/Prot_SAP_000.pdf